CLINICAL TRIAL: NCT00140361
Title: Assessing and Monitoring the Efficacy of Sulfadoxine/ Pyrimethamine (SP) and the Combination of SP Plus Artesunate for Uncomplicated Malaria Infections Among Children
Brief Title: Efficacy of Sulphadoxine-pyrimethamine and Artemisinin-containing Combination Therapy for Malaria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCID-2577; UR3/CCU018969-01
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Malaria (Uncomplicated)
Keywords: malaria; sulfadoxine-pyrimethamine; sulfadoxine-pyrimethamine plus artsunate; lumefantrine plus artemether; combination therapy
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Artesunate; Lumefantrine; Artemether

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine
Drug: sulfadoxine-pyrimethamine plus artesunate
Drug: lumefantrine plus artemether
Behavioral: Sleeping under insecticide-treated bednet

SUMMARY:
This is an ongoing monitoring activity of efficacy of sulfadoxine-pyrimethamine (SP), which is the current national treatment of choice for uncomplicated malaria in Tanzania, and a combination of SP and artesunate among children < 5 years in 3 sites in rural Tanzania.

Protocol was amended in 2004 to (1) include lumefantrine+artemether, the newly identified first-line treatment for malaria to be introduced into Tanzania in 2006; (2) on a limited basis, include adult patients; (3) extend follow-up to 28 days; (4) investigate whether treated bednets would reduce confounding by reinfection

DETAILED DESCRIPTION:
This is an ongoing monitoring activity of efficacy of sulfadoxine-pyrimethamine (SP), which is the current national treatment of choice for uncomplicated malaria in Tanzania, and a combination of SP and artesunate among children < 5 years in 3 sites in rural Tanzania.

Protocol was amended in 2004 to (1) include lumefantrine+artemether, the newly identified first-line treatment for malaria to be introduced into Tanzania in 2006; (2) on a limited basis, include adult patients; (3) extend follow-up to 28 days; (4) investigate whether treated bednets would reduce confounding by reinfection

ELIGIBILITY:
Inclusion Criteria:

Children < 5 years of age (in one site, patients of all ages are eligible).

Documented fever (axillary temperature >= 37.5oC) in the absence of another obvious cause of fever or other serious or chronic medical condition

Unmixed infection with P. falciparum of between 2,000 and 250,000 asexual parasites/mm3

Patients' or the patients' parent's or guardian's informed consent and willingness to participate in the study

Exclusion Criteria:

Any evidence of severe malaria that would require hospitalization for treatment.

Reported allergy to any antimalarial drugs, including sulfa and artemisinin drugs.

History of pregnancy or delayed menstrual period

Breastfeeding a child less than 8 weeks of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2000-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Clinical and parasitologic failure rate

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Bloland, DVM, MPVM, Principal Investigator — Centers for Disease Control and Prevention; Salim Abdulla, MD, PhD, Study Director — Ifakara Health Research and Development Centre; John R MacArthur, MD, MPH, Study Director — Centers for Disease Control and Prevention
Locations (3):
- Tanzania (3):
  - Ngere Ngere Health Center, Ngerengere, Morogoro Rural
  - Ikwiriri Health Center, Ikwiriri, Rufiji
  - Lupiro Health Center, Lupiro, Ulanga